CLINICAL TRIAL: NCT04651348
Title: A Phase I Clinical Study of Recombinant Humanized Monoclonal Antibody MIL95 Injection in the Treatment of Lymphomas and Advanced Malignant Solid Tumors
Brief Title: A Clinical Study of MIL95 in Advanced Malignancies.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL95-CT101
Record Dates: First submitted 2020-11-11; First posted 2020-12-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIL95 (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL95

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL95 — PART A :The patients confirming to the eligibility criteria will be assigned to the 4 dose groups (0.1mg/kg, 0.3mg/kg, 0.8mg/kg, 1.0mg/kg, respectively) based on the sequence of inclusion. Each patient will receive an intravenous infusion of MIL95 every week on Day 1 for a maximum of Twelve weeks.
  PART B:One recommended dose as a priming dose will be selected from 4 dose groups(0.1mg/kg、0.3mg/kg、0.8mg/kg、1.0mg/kg) based on results of PART A. Each patient will receive a priming dose of MIL95 on Day 1 Cycle 1.The patients will be assigned to the 5 maintenance dose groups (3mg/kg, 10mg/kg, 20mg/kg, 30mg/kg, 45mg/kg, respectively) based on the sequence of inclusion. The maintenance dose was given on Day 8,15,22 Cycle 1 and on Day 1,8,15,22 Cycle 2+. Each cycle was 28 days.

SUMMARY:
This study is composed of two stages: Part A initial dose escalation and Part B maintenance dose escalation. Both parts will adopt the classical 3+3 dose escalation design.

The starting dose for phase Ia part A is 0.1 mg/kg QW, followed by 3 dose cohorts (0.3mg/kg QW, 0.8mg/kg QW and 1mg/kg QW). Duration of dose limiting toxicity (DLT) observation is 14 days.

Part B will have 5 dose cohorts(3mg/kg QW, 10mg/kg QW, 20mg/kg QW 30mg/kg QW and 45mg/kg QW). DLT observation period is 28 days. The subject number for each cohort in Part B will be increased to 6 if the subject number enrolled in each cohort is less than 6.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Diagnosis of Refractory/relapsed lymphomas or solid tumor;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Life expectancy >=3 months;
5. Sufficient organ and bone marrow function;
6. At least one measurable lesion or evaluable lesion (recist v1.1 or Lugano 2014);
7. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Prior use of any anti-cancer therapy(including chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc) within 4 weeks of study start;
2. Previous exposure to any drug targeting CD47 or SIRPα;
3. Major surgery within 4 weeks prior to the first administration or expected to undergo major surgery during the study treatment;
4. Live attenuated vaccine administrated within 4 weeks before the first administration or during the study period;
5. Central nervous system metastasis;
6. History of other primary malignant tumors in 5 years;
7. Evidence of significant, uncontrolled concomitant disease;
8. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C(including HBsAg,HBcAb positive with abnormal HBV DNA or HCV RNA );
9. Active or suspected autoimmune diseases;
10. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) while participating in the study; 2) for at least 12 months after discontinuation of all study treatments;
11. Known history of hemolytic anemia;
12. Known severe allergic reaction or/and infusion reaction to monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | up to 1year after enrollment
  Percentage of Participants with AEs and SAEs assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetics:AUC | up to 1year after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics: Cmax | up to 1year after enrollment
  Maximum concentration(Cmax) of the drug after administration
Objective response rate (ORR) | up to 1year after enrollment
  To evaluate preliminary anti-tumor activity of MIL95 in subjects with advanced malignancies.ORR includes complete remission(CR) and partial remission(PR) assessed by RECIST v1.1 criteria for solid tumors and Lugano2014 criteria for lymphoma.
Duration of response (DoR) | up to 1year after enrollment
  DOR is defined as the time from the initial response (CR or PR) to the time of disease progression or death, whichever occurs first.
Progression free survival (PFS) | up to 1year after enrollment
  Defined as the time from the first day of study treatment to disease progression or death, whichever occurs first.
Immunogenicity | up to 1year after enrollment
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of MIL95.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China